CLINICAL TRIAL: NCT00877565
Title: Is Global Longitudinal Peak Systolic Strain (GLPSS) Derived From Transesophageal Echocardiography a Reliable Measure of Systolic Function? A Multicenter-Study to Compare GLPSS With Ejection Fraction Derived From Biplane Simpson´s Method on TTE and TEE in Patients Undergoing Elective Cardiac and Non-Cardiac Surgery
Brief Title: Global Longitudinal Peak Systolic Strain (GLPSS) Derived From Transesophageal Echocardiography - A Reliable Measure of Systolic Function?
Acronym: 2DSonTOEcho
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Heinz D. Tschernich, Clin. Dept. of Cardiothoracic and Vascular Anaesthesia & Intensive Medicine, Medical University of Vienna
Other Study IDs: VI_echo_01_2009
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Surgery
Keywords: LVF; Left ventricular systolic function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Systolic function is a substantial determinant of overall hemodynamics and organ function.

Therefore assessment of left ventricular systolic function (LVF) has been of central interest in Echocardiography. Ejection fraction (EF) measurement has been the gold standard echo-derived measure to describe LVF. However, EF is a blood pool derived and therefore load dependent measure.

Global longitudinal peak systolic strain average is a new parameter derived from speckle tracking tachnique. As a primarily myocardial deformation parameter it is considered to be an equivalent to EF measurement, but maybe less load dependend. The aim of the study is to investigate the reliability of GLPSS average to quantify LVF in the perioperative setting (in cardiac and non-cardiac cases).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients in the age from 19-90 years
* Cardiac and non-cardiac surgery, where intubation is indicated
* Surgical procedures with a minimum duration of 30 min
* Elective cardiac surgery on patients scheduled for correction of:

  * coronary artery disease with and without previous myocardial infarction
  * dilated cardiomyopathy; HOCM
  * disorders of the atrial or ventricular septum
  * disorders of the aortic root or the aorta
  * left and right heart valvular disease including stenotic and/or regurgitant valvular diseases.

Exclusion Criteria:

* No patient´s consent
* Contraindications for TEE (esophageal-, gastric disorders, haematologic disorders with increased bleeding incidence; ENT-surgery, surgery of the esophageus or stomach)
* Contraindications for positioning (e.g. clinical signs of acute lung edema/acute failing left or right heart, acute coronary syndrome, myocardial infarction in recent history = within 2 weeks prior to operation date)

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac and non-cardiac surgery
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-02

PRIMARY OUTCOMES:
multivariate regression-analysis | 1, 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clin. Dept. of Cardiothoracic and Vascular Anaesthesia and Intensive Medicine, Medical University of Vienna, Vienna, Austria